CLINICAL TRIAL: NCT06319040
Title: The Effect Of Addıtıonal Surgery On Muscle Strength, Proprıoceptıon And Balance In Anterıor Crucıate Lıgament Surgery
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Tugba Turk Kalkan, Principal Investigator, Medipol University
Other Study IDs: MEDİPOL MEGA 1
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Anterior Cruciate Ligament Injuries; Meniscus Lesion
Keywords: ramp lesion; muscle strength; balance; proprioception; ACL
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Lysholm Knee Score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study Group 1: 15 patients who underwent isolated ACLR
  Interventions: Other: Muscle strength measurement; Other: Knee joint proprioception; Other: Balance; Other: Fall risk test; Other: Tegner Activity Level; Other: Lysholm Knee Scoring Scale
- Study Group 2: 15 patients who underwent ACLR with additional intervention
  Interventions: Other: Muscle strength measurement; Other: Knee joint proprioception; Other: Balance; Other: Fall risk test; Other: Tegner Activity Level; Other: Lysholm Knee Scoring Scale
- Control Group: 15 healthy individuals
  Interventions: Other: Muscle strength measurement; Other: Knee joint proprioception; Other: Balance; Other: Fall risk test; Other: Tegner Activity Level; Other: Lysholm Knee Scoring Scale

INTERVENTIONS:
Other: Muscle strength measurement — Muscle strength of both legs, maximal reciprocal concentric isokinetic knee extension (quadriceps) and flexion (hamstring) at 60°/s, 90°/s and 180°/s speeds were evaluated
Other: Knee joint proprioception — Knee joint proprioception was assessed by joint position sense. Joint position sense was measured by the previously taught ability to actively find joint position (EPAB)
Other: Balance — The patients and healthy individuals participating in our study were evaluated with the General Stability Index (GSI) for general balance ability, Anterior-Posterior Stability Index (APSI) for anterior-posterior balance ability, Medial-Lateral Stability Index (MLSI) for lateral balance ability and Fall Risk Index (DRI) and Biodex Balance System (Biodex Inc., Shirley, New York, USA) for fall risk. High values obtained indicate deterioration in balance and increased risk of falling.
Other: Fall risk test — Biodex Balance System (Biodex Inc., Shirley, New York, USA) for fall risk
Other: Tegner Activity Level — Tegner Activity Level and the Turkish version of the Lysholm Knee Scoring Scale by Çelik et al. were used to subjectively determine the functional level in individuals undergoing ACL reconstruction surgery.
Other: Lysholm Knee Scoring Scale — Tegner Activity Level and the Turkish version of the Lysholm Knee Scoring Scale by Çelik et al. were used to subjectively determine the functional level in individuals undergoing ACL reconstruction surgery.

SUMMARY:
Meniscal tears and RAMP lesions are frequently seen together with ACL injuries. The aim of this study was to evaluate the effects of meniscus repair and RAMP lesion repair ACL reconstruction surgery in terms of muscle strength, proprioception, and balance. In our study, the clinical outcomes of both anterior cruciate ligament reconstruction (ACLR), medial meniscus repair (MR) and RAMP lesion repair (RR) have been compared with those of isolated ACLR.

DETAILED DESCRIPTION:
Methods:

Fifteen patients of isolated ACLR performed, 15 patients of ACLR with MR or RR performed, and 15 healthy participants were included in our study. Besides, patients to whom ACLR and additional interventions performed divide into subgroups: 7 patients with RR and 8 patients with MR. Isokinetic muscle strength, proprioception, balance, fall risk, Lysholm Knee Scoring and Tegner Activity Level scale of patients were evaluated preoperatively and at the postoperative 6th week.

The data obtained in the research were analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 22.0 program. Number, percentage, mean, and standard deviation were used as descriptive statistical methods in the evaluation of the data. The relationship between grouped variables was tested by chi-square analysis. One-way Anova test was used to compare quantitative continuous data between more than two independent groups. Scheffe test was used as a complementary post-hoc analysis to determine the differences after the Anova test. The difference between within-group measurements was analyzed with the paired-group t-test.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 40 years of age, not having had any previous knee surgery and not having any diagnosis of knee pathology, not having any musculoskeletal injury, cardiopulmonary or vestibular dysfunction that would prevent performing the tests in the study were the inclusion criteria for control group.

Exclusion Criteria:

* In addition to ACL injury, the patients with cartilage damage, knee arthrosis, misalignment in the lower extremity and additional ligament pathologies, history of previous knee surgery, any pathology in the opposite lower extremity, and additional neuromuscular diseases were excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Our study was conducted with 30 patients who were admitted to Medipol Mega University Hospital between 2018 and 2019 and were diagnosed with ACL rupture and required surgery.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
muscle strength measurement | 30 minutes
  The isokinetic system (Cybex NORM®, Humac, CA, USA) was used to assess muscle strength measurement. Subjects sat upright on the dynamometer chair with 90˚ hip flexion during measurement. The axis of rotation of the dynamometer was adjusted to align with the anatomical axis of the knee joint (lateral condyle of the femur). To prevent compensatory movements during the test, participants were fixed on both shoulders, waist, and thighs. The belt used for the tested extremity was placed 3 cm proximal to the malleolus. Both verbal and visual feedback was given for individuals to participate in the test with maximum effort

CONTACTS AND LOCATIONS:
Overall Officials: tuğba türk kalkan, MD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gulenc B, Kemah B, Yalcin S, Sayar S, Korkmaz O, Erdil M. Surgical Treatment of Meniscal RAMP Lesion. J Knee Surg. 2020 Mar;33(3):255-259. doi: 10.1055/s-0039-1677887. Epub 2019 Mar 8. PMID 30849785